CLINICAL TRIAL: NCT05462470
Title: Impact of Surgical Management for Relapse After Conversion Hepatectomy for Initially Unresectable Colorectal Liver Metastasis
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Deputy director of the department of general surgery, Fudan University
Other Study IDs: IU-CRLM
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- repeat liver surgery: repeat liver surgery for liver relapse lesions
  Interventions: Procedure: Repeat Liver Surgery
- non-repeat liver surgery: non-repeat liver surgery, just only systemic palliative chemotherapy
  Interventions: Procedure: Non-Repeat Liver Surgery

INTERVENTIONS:
Procedure: Repeat Liver Surgery — repeat liver surgery included not only hepatectomy, but also ablative treatment, including radiofrequency ablation (RFA) and microwave ablation (MWA)
  Groups: repeat liver surgery
Procedure: Non-Repeat Liver Surgery — Systemic palliative chemotherapy
  Groups: non-repeat liver surgery

SUMMARY:
For patients with initially unresectable colorectal liver metastasis (IU-CRLM) receiving effective conversion therapy, disease relapse after conversion hepatectomy is common due to the extensive tumor load. Yet, few studies have focused on the assessment and management of relapse after conversion hepatectomy for IU-CRLM. This study aimed to investigate the impact of surgical management for relapse after conversion hepatectomy in IU-CRLM.

ELIGIBILITY:
Inclusion Criteria:

* initially unresectable colorectal liver metastasis (IU-CRLM)
* received conversion therapy
* underwent conversion hepatectomy

Exclusion Criteria:

* the histologic type of CRLM was not called adenocarcinoma
* uncontrollable extrahepatic metastases, such as peritoneal, bone, brain metastasis
* history of previous hepatectomy
* the primary tumor was not resected or palliative resection
* R1 or R2 liver resection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with initially unresectable colorectal liver metastasis (IU-CRLM) underwent hepatectomy after conversion therapy
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years
  Overall survival after the first resection of liver metastatic lesions

SECONDARY OUTCOMES:
first relapse free survival | 5 years
  relapse free survival after the first resection of liver metastatic lesions
second relapse free survival | 5 years
  relapse free survival after the repeat liver surgery of liver metastatic lesions
Severe complication rate after resection of primary and metastatic lesions | 30 days after surgery
  Grade of III-V complication rate according to Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Principal Investigator — Department of General Surgery, Zhongshan Hospital, Fudan University